CLINICAL TRIAL: NCT00532571
Title: Effects of Coenzyme Q10 in PSP and CBD, A Randomized, Placebo-Controlled, Double Blind Cross Over Pilot Study
Brief Title: Effects of Coenzyme Q10 in PSP and CBD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lahey Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CoQ10 with PSP/CBD
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Progressive Supranuclear Palsy; Neurological Disorders
Keywords: CoQ10; PSP; CBD
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Nervous System Diseases | interventions — coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CoQ10

SUMMARY:
To compare the efficacy, safety and tolerability of Coenzyme Q 10 versus placebo in patients with atypical parkinsonian syndromes corticobasal degeneration (CBD) and progressive supranuclear palsy (PSP) ).

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the diagnostic criteria of PSP and CBD (above) and who were diagnosed within the past 5 years
* Age > 40
* Subjects receiving anticholinergics, amantadine, dopamine agonists, carbidopa/levodopa, eldepryl, or comtan must be on a stable dose for at least 30 days prior to baseline visit.
* Patients agreeable to participate in the study.

Exclusion Criteria:

* Prior or concurrent therapy with anticholinergics, amantadine,a dopamine agonist,carbidopa/levodopa or comtan within 30 days of the baseline visit.
* Parkinsons disease or any other atypical parkinsonism; Parkinsonism due to drugs.
* History of pallidotomy, thalamotomy, deep brain stimulation or fetal tissue transplant.
* Previous use of coenzyme Q10 within 60 days of the baseline visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Diana Apetauerova, MD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States